CLINICAL TRIAL: NCT03385694
Title: Long Term Clinical and Functional Outcome in Patients Operated on Van Ness-Borggreve Rotationplasty for Lower Limnb Bone Tumor
Brief Title: Long Term Clinical and Functional Outcome in Rotationplasty Patients
Acronym: GIROMEETING
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Mariagrazia Benedetti, MD Director Physical Medicine and Rehabilitation Unit, Istituto Ortopedico Rizzoli
Other Study IDs: 0010899
Record Dates: First submitted 2017-12-04; First posted 2017-12-28 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Disability Physical; Psychological Adaptation
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment: All the patients operated on Van Nes Rotationplasty for bone tumors at IOR and long term surviving
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — Pelvic coronal X-ray, proprioceptive test with Delos system, questionnaires administration, orthopaedic, physiatric and prosthetic assessment

SUMMARY:
Rotationplasty is a very special surgical technique. In its most frequent variant it allows, in the bone sarcomas of the distal femur, to remove all the thigh tissues including the knee joint keeping intact the innervation of the leg and the foot that are transplanted proximally after a 180 ° rotation and joined to the proximal femoral stump.

It is currently the first choice in children under the age of 6 with a bone sarcoma localized to the distal femur but also finds indication in all age groups in cases of extremely voluminous and extended to the entire thigh with the oncological need to remove in block femur, knee and all the muscular involved. The objective of the study is to obtain information about the clinical and functional status of the limb operated in long-term surviving patients. In particular in this study the problem of the possible degenerative pathology of the hip on the operated side will be addressed. Moreover the psychic and psychological well-being of this population with particular reference to gender and motherhood will be tested.

DETAILED DESCRIPTION:
30 long term survivors of rotationplasty patients at the IOR will be welcomed by the research team. They will be introduced to the aims of the research and the methodology and timing of the assessment.

The two-day agenda will be communicated to perform in a coordinated manner so that each patient performs all the exams:

* X ray pelvis
* Physiatric, orthopedic and prosthetic examination
* Proprioceptive test with Delos system
* Psychological questionnaires

ELIGIBILITY:
Inclusion Criteria:

- Rotationplasty patients operated at IOR

Exclusion Criteria:

- Disagreement of patient to participate to the study (or of part of it)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Long survivor patient operated on knee rotationplasty for bone tumors
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Hip X ray assessment | 4.12.2017 - 3.12.2018
  Pelvic frontal X-ray

SECONDARY OUTCOMES:
Physiatric Assessment | 4.12.2017 - 3.12.2018
  Muscular strenght (MMT)
Orthopaedic assessment | 4.12.2017 - 3.12.2018
  Joints ROM (degrees)
Prostheses Assessment | 4.12.2017 - 3.12.2018
  Leg lenght difference (cm)
Symptoms | 4.12.2017 - 3.12.2018
  Symptom Checklist-90
Well being | 4.12.2017 - 3.12.2018
  Psychological Well-being Scales The Italian validated version, Review of Psychiatry, 2003, 38, 3, pp.117-130) will be used. The reduced version from the 18-item test (3 items for each of the 6 dimensions of psychological well-being) will be used. Each item is assigned a score variable from 1 (= it is not my case / I do not agree) to 6 (= it is just so / perfectly agree). Some items are expressed in negative form and therefore in scoring the score assigned by the subject must be reversed. Adding the scores of the triplets you get a score for each of the 6 dimensions / subscales: autonomy, environmental control, positive relationships with others, self-acceptance, purpose in life and personal growth. Instead, the sum of the value of all 18 items gives an overall value of psychological well-being. At higher scores there is a higher level of well-being (both general and specific for each of the 6 measured dimensions).
Psychological status | 4.12.2017 - 3.12.2018
  Rosenberg Self-Esteem Scale The version translated and validated in Italian by Professor Miretta Prezza of the University of Florence (Bulletin of Applied Psychology, 1997, 223, 35-44) will be used. It measures the attitude towards oneself through 10 items, to which the subject must respond by assigning a score from 1 (strongly disagree) to 4 (strongly agree) The scores of the negative items are reversed. The total score, obtained by adding the scores of the individual items, at higher values corresponds to an attitude more positive towards oneself.
Body Image | 4.12.2017 - 3.12.2018
  Amputees Body Image Scale by James W. Breakey published in the Journal of Prosthetics and Orthotics (Volume 9, Number 2 / Spring 1997).
  It has never been translated and validated in Italian, it has been translated and adapted (to amputation + gyroplasty) for this study.
  It evaluates the disturbance in the perception of the body image on a frequency scale (from ever to ever) to 5 points ((1 = never; 5 = always) .It consists of 20 items (3 of which are expressed in 'positive' and therefore to be counted by inverting the score.) The scale gives an overall value (obtained by adding the score of all the items), which goes from 20 to 100: at higher scores there is a greater problematic in the perception of one's body image.
Balance assessment | 4.12.2017 - 3.12.2018
  Delos proprioceptive system

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benedetti MG, Okita Y, Recubini E, Mariani E, Leardini A, Manfrini M. How Much Clinical and Functional Impairment do Children Treated With Knee Rotationplasty Experience in Adulthood? Clin Orthop Relat Res. 2016 Apr;474(4):995-1004. doi: 10.1007/s11999-016-4691-9. Epub 2016 Jan 11. PMID 26754115